CLINICAL TRIAL: NCT01720316
Title: Pilot Study of Glycine Augmentation in Carriers of a Mutation in the Gene Encoding Glycine Decarboxylase
Brief Title: Neurobiology of a Mutation in Glycine Metabolism in Psychotic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Deborah L. Levy, Associate Professor, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012p001597; R21MH097470-01A1 (NIH)
Record Dates: First submitted 2012-10-30; First posted 2012-11-02 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Schizo-affective Disorder; Bipolar Disorder
Keywords: Glycine; Glycine decarboxylase; Psychosis; Mutation
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Hyperglycinemia, Nonketotic | interventions — Glycine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- glycine (Active Comparator): Glycine, up to 0.8 g/kg, administered with TID dosing for 6 weeks Double-blind
  Interventions: Drug: Glycine
- Placebo (Placebo Comparator): placebo, TID dosing, 6 weeks Double-blind
  Interventions: Drug: placebo
- glycine, open-label (Active Comparator): glycine, up to 0.8 g/kg, administered with TID dosing for 6 weeks
  Interventions: Drug: Glycine

INTERVENTIONS:
Drug: Glycine — Double-blind placebo controlled trial of glycine or placebo, followed by open-label glycine
  Arms: glycine; glycine, open-label
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of oral glycine as an augmentation strategy in two psychotic patients with a triplication (4 copies) of the gene glycine decarboxylase (GLDC). Subjects will first undergo a double-blind placebo-controlled clinical trial in which one 6-week arm will involve glycine (maximum daily dose of 0.8 g/kg, administered on a TID dosing schedule) and one 6-week arm will involve placebo. A 2-week period of no treatment will occur between treatment arms. A 6-week period of open-label glycine (maximum daily dose of 0.8 g/kg, administered on a TID dosing schedule) will follow the double-blind placebo-controlled clinical trial. Prior to the double-blind placebo-controlled clinical trial and at the end of the open-label glycine trial, the following procedures will be carried out: structural MRI (3T), Proton 1H MRS (4T), fMRI (3T), steady-state visual evoked potentials, and EEG. Positive, negative, and affective symptoms and neurocognitive function as well as plasma levels of large neutral and large and small neutral and excitatory amino acids and psychotropic drug levels will be assessed periodically. In addition, 1H MRS (4T) for 2 hours after a single oral dose of a glycine-containing drink will be assessed at baseline. Pharmaceutical grade glycine powder (Ajinomoto) or placebo will be dissolved in 20% solution and prepared by the McLean Hospital Pharmacy.

Because the results of the double-blind placebo-controlled and open-label glycine treatment arms showed substantial clinical benefit to the participants, the study has been extended to include six months of chronic open-label glycine in order to determine 1) whether the clinical benefits achieved within 6 weeks previously recur, 2) the clinical benefits are lasting, and 3) additional clinical benefits occur with longer exposure. The glycine for this extension will be provided by Letco Medical.

The investigators hypothesize that mutation carriers will have reduced endogenous brain glycine and GABA levels and increased brain glutamate and glutamine levels. Glycine administration will increase brain glycine in the two carriers, but to a lesser extent than in non-carrier family members and controls.

The investigators hypothesize reduced activation of magnocellular pathways and abnormal ERPs modulated by NMDA in mutation carriers compared with non-carrier family members and controls.

The investigators hypothesize that glycine, but not placebo, will improve positive, negative and affective symptoms as well as neurocognitive function.

The investigators also hypothesize that open-label glycine will improve clinical and cognitive functioning, will partially normalize decreased baseline glycine and GABA and increased glutamate and glutamine, and will partially normalize magnocellular pathway activation and abnormal evoked potentials.

DETAILED DESCRIPTION:
Multiple rare structural variants of relatively recent evolutionary origin are recognized as important risk factors for schizophrenia (SZ) and other neurodevelopmental disorders (e.g., autism spectrum disorders, mental retardation, epilepsy) with odds ratios as high as 7-30 (Sebat et al. 2009; Malhotra et al. 2011; Heinzen et al. 2010; Weiss et al. 2008; McCarthy et al. 2009). We have found a de novo structural rearrangement on chromosome 9p24.1 in two psychotic patients. One of the genes in this region is the gene encoding glycine decarboxylase (GLDC), which affects brain glycine metabolism. GLDC encodes the glycine decarboxylase or glycine cleavage system P-protein, which is involved in degradation of glycine in glia cells. Carriers of the GLDC triplication would be expected to have low levels of brain Gly, resulting in NMDA receptor-mediated hypofunction, which has been strongly implicated in the pathophysiology of schizophrenia (Olney & Farber, 1995; Coyle, 2006; Javitt, 2007).

There is an extensive literature on the effects of NMDA enhancing agents on positive, negative, and depressive symptoms and on neurocognitive function (see Tsai & Lin, 2010; Lin et al. 2011 for reviews). Although many studies have reported positive results in at least one symptom domain (Heresco-Levy et al. 1996, 1999, 2004; Tsai et al. 1998, 1999, 2004, 2006; Javitt et al. 2001; Goff et al. 1996; Lane et al. 2008), the results of other studies have been negative or ambiguous (Goff et al. 1999; Evins et al. 2000; Duncan et al. 2004; van Berckel et al. 1999). Factors likely to contribute to this variability include: mechanism of action of the agent, compliance, concurrent treatment with first- vs second generation antipsychotic drugs, baseline glycine blood levels, presence/absence of kynurenine pathway metabolic abnormalities (Wonodi et al. 2010; Erhardt et al. 2007) and individual differences in brain glycine uptake and metabolism (Kaufman et al. 2009; Buchanan et al. 2007). Genetic variants that impact the synthesis and breakdown of glycine, glutamate, or other modulators of NMDA receptor function are also likely to have significant effects. Although glycine augmentation has shown variable efficacy in patients unselected for having a mutation that would be expected to lower brain glycine levels, the GLDC triplication in the two carriers in this study would be expected to result in unusually low brain glycine levels, supporting its therapeutic potential as an augmentation strategy.

Thus, it is important to evaluate the therapeutic efficacy of glycine augmentation in individuals in whom there is a high prior probability of therapeutic benefit and to characterize the neurobiology of this mutation in terms of brain metabolites, brain function, and the pharmacokinetics of glycine metabolism using well-established methods (Kaufman et al. 2009; Prescot et al. 2006; Martinez et al. 2008; Butler et al. 2001; Jensen et al. 2009; Ongur et al. 2008).

ELIGIBILITY:
Inclusion Criteria:

* Triplication of glycine decarboxylase gene

Exclusion Criteria:

* Normal glycine decarboxylase copy number

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L Levy, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butler PD, Schechter I, Zemon V, Schwartz SG, Greenstein VC, Gordon J, Schroeder CE, Javitt DC. Dysfunction of early-stage visual processing in schizophrenia. Am J Psychiatry. 2001 Jul;158(7):1126-33. doi: 10.1176/appi.ajp.158.7.1126. PMID 11431235
- [Background] Buchanan RW, Javitt DC, Marder SR, Schooler NR, Gold JM, McMahon RP, Heresco-Levy U, Carpenter WT. The Cognitive and Negative Symptoms in Schizophrenia Trial (CONSIST): the efficacy of glutamatergic agents for negative symptoms and cognitive impairments. Am J Psychiatry. 2007 Oct;164(10):1593-602. doi: 10.1176/appi.ajp.2007.06081358. PMID 17898352
- [Background] Coyle JT. Glutamate and schizophrenia: beyond the dopamine hypothesis. Cell Mol Neurobiol. 2006 Jul-Aug;26(4-6):365-84. doi: 10.1007/s10571-006-9062-8. Epub 2006 Jun 14. PMID 16773445
- [Background] Duncan EJ, Szilagyi S, Schwartz MP, Bugarski-Kirola D, Kunzova A, Negi S, Stephanides M, Efferen TR, Angrist B, Peselow E, Corwin J, Gonzenbach S, Rotrosen JP. Effects of D-cycloserine on negative symptoms in schizophrenia. Schizophr Res. 2004 Dec 1;71(2-3):239-48. doi: 10.1016/j.schres.2004.03.013. PMID 15474895
- [Background] Erhardt S, Schwieler L, Nilsson L, Linderholm K, Engberg G. The kynurenic acid hypothesis of schizophrenia. Physiol Behav. 2007 Sep 10;92(1-2):203-9. doi: 10.1016/j.physbeh.2007.05.025. Epub 2007 May 21. PMID 17573079
- [Background] Evins AE, Fitzgerald SM, Wine L, Rosselli R, Goff DC. Placebo-controlled trial of glycine added to clozapine in schizophrenia. Am J Psychiatry. 2000 May;157(5):826-8. doi: 10.1176/appi.ajp.157.5.826. PMID 10784481
- [Background] Goff DC, Tsai G, Manoach DS, Flood J, Darby DG, Coyle JT. D-cycloserine added to clozapine for patients with schizophrenia. Am J Psychiatry. 1996 Dec;153(12):1628-30. doi: 10.1176/ajp.153.12.1628. PMID 8942463
- [Background] Goff DC, Henderson DC, Evins AE, Amico E. A placebo-controlled crossover trial of D-cycloserine added to clozapine in patients with schizophrenia. Biol Psychiatry. 1999 Feb 15;45(4):512-4. doi: 10.1016/s0006-3223(98)00367-9. PMID 10071726
- [Background] Heinzen EL, Radtke RA, Urban TJ, Cavalleri GL, Depondt C, Need AC, Walley NM, Nicoletti P, Ge D, Catarino CB, Duncan JS, Kasperaviciute D, Tate SK, Caboclo LO, Sander JW, Clayton L, Linney KN, Shianna KV, Gumbs CE, Smith J, Cronin KD, Maia JM, Doherty CP, Pandolfo M, Leppert D, Middleton LT, Gibson RA, Johnson MR, Matthews PM, Hosford D, Kalviainen R, Eriksson K, Kantanen AM, Dorn T, Hansen J, Kramer G, Steinhoff BJ, Wieser HG, Zumsteg D, Ortega M, Wood NW, Huxley-Jones J, Mikati M, Gallentine WB, Husain AM, Buckley PG, Stallings RL, Podgoreanu MV, Delanty N, Sisodiya SM, Goldstein DB. Rare deletions at 16p13.11 predispose to a diverse spectrum of sporadic epilepsy syndromes. Am J Hum Genet. 2010 May 14;86(5):707-18. doi: 10.1016/j.ajhg.2010.03.018. Epub 2010 Apr 15. PMID 20398883
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Horowitz A, Kelly D. Double-blind, placebo-controlled, crossover trial of glycine adjuvant therapy for treatment-resistant schizophrenia. Br J Psychiatry. 1996 Nov;169(5):610-7. doi: 10.1192/bjp.169.5.610. PMID 8932891
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Silipo G, Lichtenstein M. Efficacy of high-dose glycine in the treatment of enduring negative symptoms of schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):29-36. doi: 10.1001/archpsyc.56.1.29. PMID 9892253
- [Background] Heresco-Levy U, Ermilov M, Lichtenberg P, Bar G, Javitt DC. High-dose glycine added to olanzapine and risperidone for the treatment of schizophrenia. Biol Psychiatry. 2004 Jan 15;55(2):165-71. doi: 10.1016/s0006-3223(03)00707-8. PMID 14732596
- [Background] Javitt DC. Glutamate and schizophrenia: phencyclidine, N-methyl-D-aspartate receptors, and dopamine-glutamate interactions. Int Rev Neurobiol. 2007;78:69-108. doi: 10.1016/S0074-7742(06)78003-5. PMID 17349858
- [Background] Javitt DC, Silipo G, Cienfuegos A, Shelley AM, Bark N, Park M, Lindenmayer JP, Suckow R, Zukin SR. Adjunctive high-dose glycine in the treatment of schizophrenia. Int J Neuropsychopharmacol. 2001 Dec;4(4):385-91. doi: 10.1017/S1461145701002590. PMID 11806864
- [Background] Jensen JE, Licata SC, Ongur D, Friedman SD, Prescot AP, Henry ME, Renshaw PF. Quantification of J-resolved proton spectra in two-dimensions with LCModel using GAMMA-simulated basis sets at 4 Tesla. NMR Biomed. 2009 Aug;22(7):762-9. doi: 10.1002/nbm.1390. PMID 19388001
- [Background] Kaufman MJ, Prescot AP, Ongur D, Evins AE, Barros TL, Medeiros CL, Covell J, Wang L, Fava M, Renshaw PF. Oral glycine administration increases brain glycine/creatine ratios in men: a proton magnetic resonance spectroscopy study. Psychiatry Res. 2009 Aug 30;173(2):143-9. doi: 10.1016/j.pscychresns.2009.03.004. Epub 2009 Jun 24. PMID 19556112
- [Background] Lane HY, Liu YC, Huang CL, Chang YC, Liau CH, Perng CH, Tsai GE. Sarcosine (N-methylglycine) treatment for acute schizophrenia: a randomized, double-blind study. Biol Psychiatry. 2008 Jan 1;63(1):9-12. doi: 10.1016/j.biopsych.2007.04.038. Epub 2007 Jul 20. PMID 17659263
- [Background] Lin CH, Lane HY, Tsai GE. Glutamate signaling in the pathophysiology and therapy of schizophrenia. Pharmacol Biochem Behav. 2012 Feb;100(4):665-77. doi: 10.1016/j.pbb.2011.03.023. Epub 2011 Apr 1. PMID 21463651
- [Background] Malhotra D, McCarthy S, Michaelson JJ, Vacic V, Burdick KE, Yoon S, Cichon S, Corvin A, Gary S, Gershon ES, Gill M, Karayiorgou M, Kelsoe JR, Krastoshevsky O, Krause V, Leibenluft E, Levy DL, Makarov V, Bhandari A, Malhotra AK, McMahon FJ, Nothen MM, Potash JB, Rietschel M, Schulze TG, Sebat J. High frequencies of de novo CNVs in bipolar disorder and schizophrenia. Neuron. 2011 Dec 22;72(6):951-63. doi: 10.1016/j.neuron.2011.11.007. PMID 22196331
- [Background] Martinez A, Hillyard SA, Dias EC, Hagler DJ Jr, Butler PD, Guilfoyle DN, Jalbrzikowski M, Silipo G, Javitt DC. Magnocellular pathway impairment in schizophrenia: evidence from functional magnetic resonance imaging. J Neurosci. 2008 Jul 23;28(30):7492-500. doi: 10.1523/JNEUROSCI.1852-08.2008. PMID 18650327
- [Background] McCarthy SE, Makarov V, Kirov G, Addington AM, McClellan J, Yoon S, Perkins DO, Dickel DE, Kusenda M, Krastoshevsky O, Krause V, Kumar RA, Grozeva D, Malhotra D, Walsh T, Zackai EH, Kaplan P, Ganesh J, Krantz ID, Spinner NB, Roccanova P, Bhandari A, Pavon K, Lakshmi B, Leotta A, Kendall J, Lee YH, Vacic V, Gary S, Iakoucheva LM, Crow TJ, Christian SL, Lieberman JA, Stroup TS, Lehtimaki T, Puura K, Haldeman-Englert C, Pearl J, Goodell M, Willour VL, Derosse P, Steele J, Kassem L, Wolff J, Chitkara N, McMahon FJ, Malhotra AK, Potash JB, Schulze TG, Nothen MM, Cichon S, Rietschel M, Leibenluft E, Kustanovich V, Lajonchere CM, Sutcliffe JS, Skuse D, Gill M, Gallagher L, Mendell NR; Wellcome Trust Case Control Consortium; Craddock N, Owen MJ, O'Donovan MC, Shaikh TH, Susser E, Delisi LE, Sullivan PF, Deutsch CK, Rapoport J, Levy DL, King MC, Sebat J. Microduplications of 16p11.2 are associated with schizophrenia. Nat Genet. 2009 Nov;41(11):1223-7. doi: 10.1038/ng.474. Epub 2009 Oct 25. PMID 19855392
- [Background] Olney JW, Farber NB. Glutamate receptor dysfunction and schizophrenia. Arch Gen Psychiatry. 1995 Dec;52(12):998-1007. doi: 10.1001/archpsyc.1995.03950240016004. PMID 7492260
- [Background] Ongur D, Jensen JE, Prescot AP, Stork C, Lundy M, Cohen BM, Renshaw PF. Abnormal glutamatergic neurotransmission and neuronal-glial interactions in acute mania. Biol Psychiatry. 2008 Oct 15;64(8):718-726. doi: 10.1016/j.biopsych.2008.05.014. Epub 2008 Jul 7. PMID 18602089
- [Background] Prescot AP, de B Frederick B, Wang L, Brown J, Jensen JE, Kaufman MJ, Renshaw PF. In vivo detection of brain glycine with echo-time-averaged (1)H magnetic resonance spectroscopy at 4.0 T. Magn Reson Med. 2006 Mar;55(3):681-6. doi: 10.1002/mrm.20807. PMID 16453318
- [Background] Sebat J, Levy DL, McCarthy SE. Rare structural variants in schizophrenia: one disorder, multiple mutations; one mutation, multiple disorders. Trends Genet. 2009 Dec;25(12):528-35. doi: 10.1016/j.tig.2009.10.004. Epub 2009 Oct 31. PMID 19883952
- [Background] Tsai GE, Lin PY. Strategies to enhance N-methyl-D-aspartate receptor-mediated neurotransmission in schizophrenia, a critical review and meta-analysis. Curr Pharm Des. 2010;16(5):522-37. doi: 10.2174/138161210790361452. PMID 19909229
- [Background] Tsai GE, Yang P, Chung LC, Tsai IC, Tsai CW, Coyle JT. D-serine added to clozapine for the treatment of schizophrenia. Am J Psychiatry. 1999 Nov;156(11):1822-5. doi: 10.1176/ajp.156.11.1822. PMID 10553752
- [Background] Tsai G, Yang P, Chung LC, Lange N, Coyle JT. D-serine added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 1998 Dec 1;44(11):1081-9. doi: 10.1016/s0006-3223(98)00279-0. PMID 9836012
- [Background] Tsai G, Lane HY, Yang P, Chong MY, Lange N. Glycine transporter I inhibitor, N-methylglycine (sarcosine), added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 2004 Mar 1;55(5):452-6. doi: 10.1016/j.biopsych.2003.09.012. PMID 15023571
- [Background] Tsai GE, Yang P, Chang YC, Chong MY. D-alanine added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 2006 Feb 1;59(3):230-4. doi: 10.1016/j.biopsych.2005.06.032. Epub 2005 Sep 9. PMID 16154544
- [Background] van Berckel BN, Evenblij CN, van Loon BJ, Maas MF, van der Geld MA, Wynne HJ, van Ree JM, Kahn RS. D-cycloserine increases positive symptoms in chronic schizophrenic patients when administered in addition to antipsychotics: a double-blind, parallel, placebo-controlled study. Neuropsychopharmacology. 1999 Aug;21(2):203-10. doi: 10.1016/S0893-133X(99)00014-7. PMID 10432468
- [Background] Weiss LA, Shen Y, Korn JM, Arking DE, Miller DT, Fossdal R, Saemundsen E, Stefansson H, Ferreira MA, Green T, Platt OS, Ruderfer DM, Walsh CA, Altshuler D, Chakravarti A, Tanzi RE, Stefansson K, Santangelo SL, Gusella JF, Sklar P, Wu BL, Daly MJ; Autism Consortium. Association between microdeletion and microduplication at 16p11.2 and autism. N Engl J Med. 2008 Feb 14;358(7):667-75. doi: 10.1056/NEJMoa075974. Epub 2008 Jan 9. PMID 18184952
- [Background] Wonodi I, Schwarcz R. Cortical kynurenine pathway metabolism: a novel target for cognitive enhancement in Schizophrenia. Schizophr Bull. 2010 Mar;36(2):211-8. doi: 10.1093/schbul/sbq002. Epub 2010 Feb 10. PMID 20147364
- [Derived] Bodkin JA, Coleman MJ, Godfrey LJ, Carvalho CMB, Morgan CJ, Suckow RF, Anderson T, Ongur D, Kaufman MJ, Lewandowski KE, Siegel AJ, Waldstreicher E, Grochowski CM, Javitt DC, Rujescu D, Hebbring S, Weinshilboum R, Rodriguez SB, Kirchhoff C, Visscher T, Vuckovic A, Fialkowski A, McCarthy S, Malhotra D, Sebat J, Goff DC, Hudson JI, Lupski JR, Coyle JT, Rudolph U, Levy DL. Targeted Treatment of Individuals With Psychosis Carrying a Copy Number Variant Containing a Genomic Triplication of the Glycine Decarboxylase Gene. Biol Psychiatry. 2019 Oct 1;86(7):523-535. doi: 10.1016/j.biopsych.2019.04.031. Epub 2019 May 9. PMID 31279534

RESULTS

PARTICIPANT FLOW:
Groups:
- Glycine, Then Placebo: One participant received glycine powder, up to 0.8 g/kg, administered with TID dosing for 6 weeks, then the participant received placebo TID dosing for 6 weeks, then the participant received open-label glycine for 6 weeks.
- Placebo, Then Glycine: One participant received placebo administered with TID dosing for 6 weeks, then the participant received glycine powder, up to 0.8 g/kg, TID dosing for 6 weeks, then the participant received open-label glycine for 6 weeks.
Period: Double-Blind Glycine Placebo Crossover
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Open-label Glycine
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Glycine, Then Placebo: One participant received glycine powder, up to 0.8 g/kg, administered with TID dosing for 6 weeks, then the participant received placebo TID dosing for 6 weeks, then open-label glycine for 6 weeks.
- Placebo, Then Glycine: One participant received placebo administered with TID dosing for 6 weeks, then the participant received glycine powder, up to 0.8 g/kg, TID dosing for 6 weeks, then open-label glycine for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] — age at beginning of study
  years
    age | 59 [NA to NA] — Single participant in each arm | 32 [NA to NA] — Single participant in each arm | 45.5 [32 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Symptom Scores at Baseline and at 2 Weeks, 4 Weeks, and 6 Weeks During Intervention 1 (Glycine or Placebo), Intervention 2 (Glycine or Placebo), and During Open-label Glycine
Description: Positive and Negative Symptom Scale (PANSS) measures positive and negative symptoms of schizophrenia. The sum of ratings for seven positive symptoms are measured on a scale from 7-49 with 7 meaning no symptoms and 49 meaning severe symptoms.
Time Frame: baseline and at 2 weeks, 4 weeks, and 6 weeks within each treatment period and after each treatment period
Measure: Number; unit: units on a scale
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Number analyzed (Participants) | 1 | 1
units on a scale
  Positive symptoms at baseline | 13 | 19
  Positive symptoms at 2 weeks intervention 1 | 12 | 20
  Positive symptoms at 4 weeks intervention 1 | 9 | 19
  Positive symptoms at 6 weeks intervention 1 | 8 | 13
  Positive symptoms, end of washout1 | 7 | 13
  Positive symptoms at 2 weeks intervention 2 | 12 | 12
  Positive symptoms at 4 weeks intervention 2 | 11 | 10
  Positive symptoms at 6 weeks intervention 2 | 14 | 11
  Positive symptoms, end of washout2 | 14 | 11
  Positive symptoms at 2 weeks open label | 9 | 8
  Positive symptoms at 4 weeks open label | 9 | 7
  Positive symptoms at 6 weeks open label | 7 | 8
  Positive symptoms, end of washout3 | 7 | 8

2. Primary Outcome: Neurocognitive Function at Baseline, During Glycine Treatment, During Placebo Treatment and During Open-label Glycine
Description: Scores on each of 8 domains of cognitive function (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning/problem solving, social cognition, overall composite). Scores are T scores ranging from 0-100, with 50 representing the mean for a population based on a normal distribution; standard deviation of 10. Only overall composite score is entered.
Time Frame: At baseline, during glycine treatment, during placebo treatment and during open-label glycine
Population: Data provided for each participant separately.
Measure: Number; unit: units on a scale
Groups:
- Baseline: Composite Score at Baseline
- Composite Score on Glycine, Double-blind: Glycine, up to 0.8 g/kg, administered with TID dosing for 6 weeks Double-blind
  Glycine: Double-blind placebo controlled trial of glycine or placebo, followed by open-label glycine
- Composite Score on Placebo: placebo, TID dosing, 6 weeks Double-blind
  placebo
- Composite Score on Glycine, Open-label: glycine, up to 0.8 g/kg, administered with TID dosing for 6 weeks
  Glycine: Double-blind placebo controlled trial of glycine or placebo, followed by open-label glycine
Arm/Group | Baseline | Composite Score on Glycine, Double-blind | Composite Score on Placebo | Composite Score on Glycine, Open-label
Number analyzed (Participants) | 2 | 2 | 2 | 2
units on a scale
  Participant 1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 1 | 45 | 52 | 52 | 49
  Participant 2: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 2 | 48 | 52 | 55 | 46

3. Primary Outcome: Glycine Plasma Amino Acid Levels at Baseline, During Glycine Treatment, During Placebo Treatment and During Open-label Glycine
Description: Plasma glycine levels; normal range is 122-467 nM/mL
Time Frame: At baseline, during glycine treatment, during placebo treatment and during open-label glycine
Measure: Number; unit: nM/mL
Groups:
- Glycine Then Placebo: Glycine, up to 0.8 g/kg, administered with TID dosing for 6 weeks Double-blind
  Glycine: Double-blind placebo controlled trial of glycine or placebo, followed by open-label glycine
- Placebo Then Glycine: placebo, TID dosing, 6 weeks Double-blind
  placebo
Arm/Group | Glycine Then Placebo | Placebo Then Glycine
Number analyzed (Participants) | 1 | 1
nM/mL
  Baseline | 216 | 271
  Glycine double-blind | 410 | 761
  Placebo | 194 | 347
  Glycine open-label | 516 | 634

4. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Scores at Baseline and at 2 Weeks, 4 Weeks, and 6 Weeks Positive and Negative Symptom Scores at Baseline and at 2, 4, and 6 Weeks During Intervention 1, Intervention 2, and During Open-label Glycine
Description: Total BPRS score measures severity of 18 psychiatric symptoms. Each symptom is scored 1-7 with the total score ranging from 18-126. 18 means no symptoms and 126 means very severe symptoms.
Time Frame: baseline and at 2 weeks, 4 weeks, and 6 weeks within and after each treatment period
Measure: Number; unit: units on a scale
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Number analyzed (Participants) | 1 | 1
units on a scale
  BPRS at baseline | 39 | 46
  BPRS at 2 weeks intervention 1 | 38 | 38
  BPRS at 4 weeks intervention 1 | 32 | 39
  BPRS at 6 weeks intervention 1 | 21 | 28
  BPRS, end of washout1 | 22 | 34
  BPRS at 2 weeks intervention 2 | 37 | 32
  BPRS at 4 weeks intervention 2 | 31 | 20
  BPRS at 6 weeks intervention 2 | 37 | 23
  BPRS, end of washout2 | 32 | 24
  BPRS at 2 weeks open label | 23 | 20
  BPRS at 4 weeks open label | 22 | 18
  BPRS at 6 weeks open label | 21 | 19
  BPRS, end of washout3 | 19 | 23

5. Primary Outcome: Clinical Global Impression (CGI) Severity Scores at Baseline and at 2 Weeks, 4 Weeks, and 6 Weeks Within Each Treatment Period
Description: Clinical Global Impression (CGI) severity scores measure severity of mental illness on a scale of 1-7 where 1 means normal, not at all ill, 2 means borderline mentally ill, 3 means mildly ill, 4 means moderately ill, 5 means markedly ill, 6 means severely ill and 7 means among the most extremely ill patients.
Time Frame: CGI at baseline and at 2 weeks, 4 weeks, and 6 weeks per treatment period
Measure: Number; unit: units on a scale
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Number analyzed (Participants) | 1 | 1
units on a scale
  CGI severity score at baseline | 4 | 4
  CGI severity score at 2 weeks intervention 1 | 4 | 4
  CGI severity score at 4 weeks intervention 1 | 3 | 4
  CGI severity score at 6 weeks intervention 1 | 2 | 4
  CGI severity score, end of washout1 | 2 | 4
  CGI severity score at 2 weeks intervention 2 | 4 | 4
  CGI severity score at 4 weeks intervention 2 | 4 | 4
  CGI severity score at 6 weeks intervention 2 | 4 | 3
  CGI severity score, end of washout2 | 4 | 3
  CGI severity score at 2 weeks open label | 3 | 3
  CGI severity score at 4 weeks open label | 3 | 3
  CGI severity score at 6 weeks open label | 2 | 2
  CGI severity score, end of washout3 | 2 | 2

6. Primary Outcome: Clinical Global Impression (CGI) Therapeutic Effect Scores at 2 Weeks, 4 Weeks, and 6 Weeks Within Each Treatment Period
Description: Clinical Global Impression (CGI) therapeutic effect scores measure degree of improvement as marked (1), moderate (5), minimal (9) or unchanged/worse (13).
Time Frame: at 2 weeks, 4 weeks, and 6 weeks within each treatment period
Measure: Number; unit: score
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Number analyzed (Participants) | 1 | 1
score
  CGI therapeutic effect at 2 weeks intervention 1 | 13 | 5
  CGI therapeutic effect at 4 weeks intervention 1 | 5 | 5
  CGI therapeutic effect at 6 weeks intervention 1 | 5 | 5
  CGI therapeutic effect, end of washout1 | 5 | 5
  CGI therapeutic effect at 2 weeks intervention 2 | 13 | 13
  CGI therapeutic effect at 4 weeks intervention 2 | 13 | 5
  CGI therapeutic effect at 6 weeks intervention 2 | 13 | 5
  CGI therapeutic effect, end of washout2 | 13 | 5
  CGI therapeutic effect at 2 weeks open label | 5 | 1
  CGI therapeutic effect at 4 weeks open label | 5 | 1
  CGI therapeutic effect at 6 weeks open label | 1 | 1
  CGI therapeutic effect, end of washout3 | 1 | 1

7. Primary Outcome: Mania Symptom Scores at Baseline and at 2 Weeks, 4 Weeks, and 6 Weeks Within Each Treatment Period
Description: Young Mania Rating Scale (YMRS) measures severity of manic symptoms. The sum of ratings for 7 symptoms of mania is measured on a scale from 0-4 and the sum of 4 symptoms of mania is measured on a scale from 0-8 to yield a total score ranging from 0-60, with 0 meaning no manic symptoms and 60 meaning severe manic symptoms.
Time Frame: baseline and at 2 weeks, 4 weeks, and 6 weeks within each treatment period
Measure: Number; unit: units on a scale
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Number analyzed (Participants) | 1 | 1
units on a scale
  Manic symptoms at baseline | 4 | 7
  Manic symptoms at 2 weeks intervention 1 | 1 | 7
  Manic symptoms at 4 weeks intervention 1 | 0 | 6
  Manic symptoms at 6 weeks intervention 1 | 0 | 0
  Manic symptoms, end of washout1 | 0 | 0
  Manic symptoms at 2 weeks intervention 2 | 17 | 0
  Manic symptoms at 4 weeks intervention 2 | 0 | 0
  Manic symptoms at 6 weeks intervention 2 | 2 | 0
  Manic symptoms, end of washout2 | 2 | 0
  Manic symptoms at 2 weeks open label | 1 | 0
  Manic symptoms at 4 weeks open label | 0 | 0
  Manic symptoms at 6 weeks open label | 0 | 0
  Manic symptoms, end of washout3 | 0 | 0

8. Primary Outcome: Depression Symptom Scores at Baseline and at 2 Weeks, 4 Weeks, and 6 Weeks Within Each Treatment Period
Description: Hamilton Depression Scale measures severity of depression symptoms. The sum of ratings for 9 depression symptoms are measured on a scale from 0-2 with 0 meaning no symptoms and 2 meaning some level of severity of that specific symptom. The rating for 1 depression symptom is measured on a scale from 0-3 with 0 meaning no symptoms and 3 meaning a severe level of that specific symptom. The sum of ratings for 11 depression symptoms are measured on a scale from 0-4 with 0 meaning no symptoms and 4 meaning a severe level of that specific symptom. The three sums are added to produce an overall depression rating scale score ranging from 0-65.
Time Frame: baseline and at 2 weeks, 4 weeks, and 6 weeks within each treatment period
Measure: Number; unit: units on a scale
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Number analyzed (Participants) | 1 | 1
units on a scale
  Depression symptoms at baseline | 18 | 12
  Depression symptoms at 2 weeks intervention 1 | 17 | 5
  Depression symptoms at 4 weeks intervention 1 | 11 | 5
  Depression symptoms at 6 weeks intervention 1 | 3 | 0
  Depression symptoms, end of washout1 | 1 | 3
  Depression symptoms at 2 weeks intervention 2 | 19 | 3
  Depression symptoms at 4 weeks intervention 2 | 5 | 2
  Depression symptoms at 6 weeks intervention 2 | 7 | 1
  Depression symptoms, end of washout2 | 3 | 1
  Depression symptoms at 2 weeks open label | 2 | 1
  Depression symptoms at 4 weeks open label | 2 | 1
  Depression symptoms at 6 weeks open label | 1 | 1
  Depression symptoms, end of washout3 | 2 | 0

9. Secondary Outcome: Brain Glycine/CR Ratio
Description: magnetic resonance spectroscopy: glycine/creatine ratio. Participants were assessed at 1) BASELINE PRE-GLYCINE TREATMENT: pre-glycine challenge drink, 60 minutes post challenge drink, 80 minutes post challenge drink, 100 minutes post challenge drink, and 120 minutes post challenge drink (0.4 g/kg up to max of 30 g); and 2) IN WEEK 6 OF OPEN-LABEL GLYCINE TREATMENT: pre-glycine dose, and 60 minutes, 80 minutes, 100 minutes and 120 minutes post daily dose of glycine. Measured in posterior occipital cortex
Time Frame: baseline (pre-challenge, 60, 80, 100, 120 minutes post-challenge), and week 6 of glycine (pre-dose and 60, 80, 100, 120 minutes post-dose
Measure: Number; unit: ratio
Groups:
- Subject1: Brain Glycine/CR Ratio at Baseline/Week 6 of Glycine: Brain glycine/CR ratio at baseline and week 6 of glycine for one participant: Subject 1
- Subject 2:Brain Glycine/CR Ratio at Baseline/Week 6 of Glycine: Brain glycine/CR ratio at baseline and week 6 of glycine for one participant
Arm/Group | Subject1: Brain Glycine/CR Ratio at Baseline/Week 6 of Glycine | Subject 2:Brain Glycine/CR Ratio at Baseline/Week 6 of Glycine
Number analyzed (Participants) | 1 | 1
ratio
  Baseline - pre-challenge drink | 0.2558 | 0.5691
  Baseline 60 minutes post challenge drink | 0.6157 | 0.3918
  Baseline 80 minutes post challenge drink | 0.6631 | 0.6428
  Baseline 100 minutes post challenge drink | 0.5938 | 0.6363
  Baseline 120 minutes post challenge drink | 0.6953 | 0.9559
  Week 6 of glycine - pre-glycine dose | 0.6573 | 0.3235
  Week 6 of glycine - 60 minutes post glycine dose | 0.2983 | 0.3807
  Week 6 of glycine - 80 minutes post glycine dose | 0.4577 | 0.5591
  Week 6 of glycine - 100 minutes post glycine dose | 0.5751 | 0.4142
  Week 6 of glycine - 120 minutes post glycine dose | 0.3842 | 0.3545

10. Secondary Outcome: Brain Glutamate Metabolite Levels (Glutamate/Creatine Ratio: Glu/Cr) at 1) BASELINE - Pre-glycine Treatment and 2) IN WEEK 6 OF GLYCINE TREATMENT
Description: magnetic resonance spectroscopy - glutamate metabolite level. Participants were assessed 1) pre-glycine treatment and in week 6 of open-label glycine treatment. Measured in posterior occipital cortex.
Time Frame: baseline and week 6 of glycine
Measure: Number; unit: ratio
Groups:
- Subject1: Brain Glutamate/CR Ratio- Baseline/Week 6 of Glycine: Brain glutamate/CR ratio at baseline and week 6 of glycine for one participant: Subject 1
- Subject2: Brain Glutamate/CR Ratio- Baseline/Week 6 of Glycine: Brain glutamate/CR ratio at baseline and week 6 of glycine for one participant: Subject 2
Arm/Group | Subject1: Brain Glutamate/CR Ratio- Baseline/Week 6 of Glycine | Subject2: Brain Glutamate/CR Ratio- Baseline/Week 6 of Glycine
Number analyzed (Participants) | 1 | 1
ratio
  Baseline brain glutamate/Cr ratio | 0.98 | 2.053
  Week 6 brain glutamate/Cr ratio | 0.84 | 1.13

11. Secondary Outcome: Brain GABA Metabolite Levels (GABA/Creatine Ratio: GABA/Cr) at 1) BASELINE - Pre-glycine Treatment and 2) IN WEEK 6 OF GLYCINE TREATMENT
Description: Magnetic resonance spectroscopy GABA/Cr. Participants were assessed 1) pre-glycine treatment (baseline) and 2) in week 6 of open-label glycine treatment measured in posterior occipital cortex.
Time Frame: Baseline and week 6 of glycine
Measure: Number; unit: ratio
Groups:
- Subject1: Brain GABA/CR Ratio- Baseline/Week 6 of Glycine: Brain GABA/CR ratio at baseline and week 6 of glycine for one participant: Subject 1
- Subject2: Brain GABA/CR Ratio- Baseline/Week 6 of Glycine: Brain GABA/CR ratio at baseline and week 6 of glycine for one participant: Subject 2
Arm/Group | Subject1: Brain GABA/CR Ratio- Baseline/Week 6 of Glycine | Subject2: Brain GABA/CR Ratio- Baseline/Week 6 of Glycine
Number analyzed (Participants) | 1 | 1
ratio
  Baseline GABA/Cr | 0.16 | 0.27
  Week 6 of glycine tx GABA/Cr | 0.22 | 0.24

12. Secondary Outcome: Auditory Evoked Potentials in Latency (Msec) at BASELINE - Pre-glycine Treatment and 2) IN WEEK 6 OF TREATMENT WITH GLYCINE
Description: Auditory evoked potentials latency: P300 at fz, cz, and pz); N100 at fz and cz); P200 at fz and cz. Participants were assessed at baseline and in week of open-label glycine treatment.
Time Frame: Recordings at baseline and week 6 of glycine
Population: Only one subject received these procedures because normal hearing is required.
Measure: Number; unit: msec
Groups:
- Auditory ERPs Latency (ms) Baseline: Subject 1: Subject1: Auditory ERPs (latency) baseline
- Auditory ERPs Latency (ms) 6 Weeks of Glycine: Subject 1: Subject1: Auditory ERPs (latency) week 6 of glycine
- Auditory ERPs Latency (ms) Baseline: Subject 2: Subject2: Auditory ERPs (latency) baseline
- Auditory ERPs Latency (ms) 6 Weeks of Glycine: Subject 2: Subject2: Auditory ERPs (latency) week 6 of glycine
Arm/Group | Auditory ERPs Latency (ms) Baseline: Subject 1 | Auditory ERPs Latency (ms) 6 Weeks of Glycine: Subject 1 | Auditory ERPs Latency (ms) Baseline: Subject 2 | Auditory ERPs Latency (ms) 6 Weeks of Glycine: Subject 2
Number analyzed (Participants) | 0 | 0 | 1 | 1
msec
  P300 latency at fz |  |  | 279.3 | 300.78
  P300 latency at cz |  |  | 279.3 | 293
  P300 latency at pz |  |  | 279.3 | 294.92
  N100 latency at fz |  |  | 97.66 | 94
  N100 latency at cz |  |  | 91.8 | 94
  P200 latency at fz |  |  | 197.27 | 205
  P200 latency at cz |  |  | 193.4 | 203

13. Secondary Outcome: Change in Magnocellular Pathway Function on Glycine Compared With Baseline. No Data Were Collected.
Description: functional magnetic resonance imaging
Time Frame: 6 weeks per treatment arm
Population: Data not collected.
Groups:
- Glycine: Glycine powder, up to 0.8 g/kg, administered with TID dosing for 6 weeks
  glycine powder: Double-blind placebo controlled trial of glycine or placebo, followed by open-label glycine
- Placebo: placebo, TID dosing, 6 weeks
  placebo
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Auditory Evoked Potentials in Amplitude (Degrees Measured in Microvolts) at 1) BASELINE - Pre-glycine Treatment and 2) IN WEEK 6 OF GLYCINE TREATMENT
Description: Auditory evoked potentials amplitude: P300 at fz, cz, and pz; N100 at fz and cz; P200 at fz and cz; P50 S1 and S2 amplitude; mismatch negativity (MMN) at fz and cz. Participants were assessed at baseline and in week 6 of open-label glycine treatment.
Time Frame: Recordings at baseline and week 6 of glycine
Population: Only one subject received these procedures because normal hearing is required.
Measure: Number; unit: microvolts
Groups:
- Auditory ERPs Amplitude (Deg) Baseline: Subject 1: Subject1: Auditory ERPs (amplitude) baseline
- Auditory ERPs Amplitude (Deg) 6 Weeks of Glycine: Subject 1: Subject1: Auditory ERPs (amplitude) week 6 of glycine
- Auditory ERPs Amplitude (Deg) Baseline: Subject 2: Subject2: Auditory ERPs (amplitude) baseline
- Auditory ERPs Amplitude (Deg) 6 Weeks of Glycine: Subject 2: Subject2: Auditory ERPs (amplitude) week 6 of glycine
Arm/Group | Auditory ERPs Amplitude (Deg) Baseline: Subject 1 | Auditory ERPs Amplitude (Deg) 6 Weeks of Glycine: Subject 1 | Auditory ERPs Amplitude (Deg) Baseline: Subject 2 | Auditory ERPs Amplitude (Deg) 6 Weeks of Glycine: Subject 2
Number analyzed (Participants) | 0 | 0 | 1 | 1
microvolts
  P300 amplitude at fz |  |  | -0.635 | 3.74
  P300 amplitude at cz |  |  | 6.53 | 6.6
  P300 amplitude at pz |  |  | 5.34 | 5.57
  N100 amplitude at fz |  |  | -3.93 | -4.71
  N100 amplitude at cz |  |  | -3.62 | -3.89
  P200 amplitude at fz |  |  | 1.662 | 6.29
  P200 amplitude at cz |  |  | 6.59 | 7.8
  P50 S1 amplitude |  |  | 2.76 | 2.2
  P50 S2 amplitude |  |  | 1.23 | 0.78
  MMN amplitude at fz |  |  | -3.356 | -1.004
  MMN amplitude at cz |  |  | -4.13 | -1.322

15. Secondary Outcome: Auditory Evoked Potentials in Gammas Oscillations (the Power Spectrum is Measured in Microvolts Squared) at 1) BASELINE - Pre-glycine Treatment and 2) IN WEEK 6 OF GLYCINE TREATMENT
Description: Auditory evoked potentials gamma: G40 hz phase locking at fz and cz; G20 hz phase locking response at fz and cz G30 hz phase locking response at fz and cz. Participants were assessed at baseline and in week 6 of open-label glycine treatment.
Time Frame: Recordings at baseline and week 6 of glycine
Population: Only one subject received these procedures because normal hearing is required.
Measure: Number; unit: microvolts squared
Groups:
- Auditory ERPs Gamma Baseline: Subject 1: Subject1: Auditory ERPs (gamma phase locking) baseline
- Auditory ERPs Gamma 6 Weeks of Glycine: Subject 1: Subject1: Auditory ERPs (gamma phase locking) week 6 of glycine
- Auditory ERPs Gamma Baseline: Subject 2: Subject2: Auditory ERPs (gamma phase locking) baseline
- Auditory ERPs Gamma 6 Weeks of Glycine: Subject 2: Subject2: Auditory ERPs (gamma phase locking) week 6 of glycine
Arm/Group | Auditory ERPs Gamma Baseline: Subject 1 | Auditory ERPs Gamma 6 Weeks of Glycine: Subject 1 | Auditory ERPs Gamma Baseline: Subject 2 | Auditory ERPs Gamma 6 Weeks of Glycine: Subject 2
Number analyzed (Participants) | 0 | 0 | 1 | 1
microvolts squared
  G40 fz |  |  | 0.135 | 0.255
  G40 cz |  |  | 0.168 | 0.29
  G20 fz |  |  | 0.023 | 0.107
  G20 cz |  |  | 0.03 | 0.108
  G30 fz |  |  | 0.19 | 0.177
  G30 cz |  |  | 0.163 | 0.242

16. Secondary Outcome: Auditory Evoked Potentials - P50 Ratio (P50 S2/P50 S1 Amplitude) at 1) BASELINE - Pre-glycine Treatment and 2) IN WEEK 6 OF GLYCINE TREATMENT
Description: Auditory evoked potentials amplitude: P50 ratio (S2/S1). Participants were assessed at baseline and in week 6 of open-label glycine treatment.
Time Frame: Recordings at baseline and week 6 of glycine
Population: Only one subject received these procedures because normal hearing is required.
Measure: Number; unit: ratio
Arm/Group | Auditory ERPs Amplitude (Deg) Baseline: Subject 1 | Auditory ERPs Amplitude (Deg) 6 Weeks of Glycine: Subject 1 | Auditory ERPs Amplitude (Deg) Baseline: Subject 2 | Auditory ERPs Amplitude (Deg) 6 Weeks of Glycine: Subject 2
Number analyzed (Participants) | 0 | 0 | 1 | 1
ratio |  |  | 44.51 | 35.67

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Glycine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycine (N=2) | Placebo (N=2)
nausea (Gastrointestinal disorders) | 2 | 0
vomiting (Gastrointestinal disorders) | 2 | 0
diarrhea (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2012-11-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT01720316/ICF_000.pdf
  • Statistical Analysis Plan (2012-10-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT01720316/SAP_001.pdf
  • Study Protocol (2012-10-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT01720316/Prot_002.pdf